CLINICAL TRIAL: NCT05205486
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of a Single 3 Gram Dose of Cefazolin in Adult Subjects Weighing >= 120 kg Scheduled for Surgery
Brief Title: Pharmacokinetics and Safety of Cefazolin 3gm DUPLEX in Adults
Acronym: 3gCefPK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: US-G-H-2101
Record Dates: First submitted 2021-10-11; First posted 2022-01-25 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Infections
Keywords: Cephalosporin; antibiotic; infection control; surgical prophylaxis
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized pharmacokinetic study. All subjects will be receiving the same study treatment, thus blinding is unnecessary.
Masking Description: This is an open-label, non-randomized pharmacokinetic study. All subjects will be receiving the same study treatment, thus masking is unnecessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cefazolin 3gm Injection (Experimental): Study drug will be administrated as an infusion over 30 minutes starting approximately 0.5 hours before surgery begins and following institutional guidelines on Day 1 (day of surgery). All subjects will have five (5) individual whole blood samples (4 mL each) collected for the estimation of cefazolin concentration in plasma at the following times after the start of the infusion: 0.5 (+/-10 min) end of infusion, 1 h (+/-15 min), 2 h (+/-15 min), 4 h (+/-15 min), and 8 h (+/-15 min).
  Interventions: Drug: Cefazolin 3gm for Injection USP and Dextrose Injection USP

INTERVENTIONS:
Drug: Cefazolin 3gm for Injection USP and Dextrose Injection USP — Cefazolin 3gm for Injection USP and Dextrose Injection USP in the DUPLEX® Drug Delivery System. Administration will occur once as a 30 minute IV infusion prior to surgery in adult subjects weighing >/= 120 kg
  Other Names: Cefazolin 3gm in DUPLEX (50ml)

SUMMARY:
This study is designed to evaluate the pharmacokinetics (PK) of a single 3 gm dose of cefazolin from a DUPLEX container, in adult subjects (weighing >/= 120 kg) scheduled for surgery. Cefazolin will be administered as a 30-minute intravenous (IV) infusion, per cefazolin Package Insert. Five PK samples per subject will be obtained up to 8 hours after dosing. These data will then be assessed by the validated Cefazolin PK Model to verify there are no significant PK changes within this study population.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose, multiple-center, study to determine the pharmacokinetics of a single 3 g dose of cefazolin administered as a 30 minute IV infusion prior to surgery in adult subjects weighing >/= 120 kg. Adult subjects will be enrolled in order to ensure at least 12 subjects complete the study. Enrollment will be competitive across the study sites. All subjects will have Screening and baseline evaluations performed to ensure their eligibility for the study The Screening Period is up to 30 days before administration of study drug on Day 1.

Study drug will be administrated as an infusion over 30 minutes starting approximately 0.5 hours before surgery begins and following institutional guidelines on Day 1 (day of surgery). Planned surgical procedures may be performed outpatient or inpatient and are expected to last no longer than 3 hours.

If the surgery is extended unexpectedly beyond the 3-hour limit, additional doses of study drug are permitted according to institutional guidelines. PK blood sample collection will continue after the administration of an additional dose of cefazolin. Safety in this population will also be assessed.

All subjects will have five (5) individual whole blood samples (4 mL each) collected for the estimation of cefazolin concentration in plasma at the following times after the start of the infusion: 0.5 (+/-10 min) end of infusion, 1 h (+/-15 min), 2 h (+/-15 min), 4 h (+/-15 min) and 8 h (+/-15 min).

Safety will be assessed by monitoring adverse events (AEs), physical examination, vital signs, and clinical laboratory tests. A follow-up visit will be performed on Day 8 (+/-1 day) for safety assessments.

A subject is considered a study completer if he/she has completed all study related procedures through the end of surgery and the required PK sample collections. It is highly preferred that the subjects also participate in the Day 8 (+/-1 day) Safety Follow-up. For subjects who withdraw or are withdrawn before study completion of the study, every effort will be made to perform all Safety Follow up procedures.

Any subject who withdraws or is withdrawn before collection of at least 4 of the 5 PK samples will not be consider as a PK completer. If necessary, additional subjects must be enrolled to ensure that there are at least 12 PK completers.

On Day 8 (+/-1 day), a Safety follow-up will be conducted. If this is an in-person visit, the following will be performed: vital signs, clinical laboratory tests, examination of the infusion site, review of AEs and concomitant medication. If an in-person visit is not possible, every effort will be made to contact the subject by phone and the subjects will be asked about any AEs and concomitant medication they may have taken.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged >/= 18 years;
2. Must weigh >/= 120 kg
3. Able to understand and sign the Informed Consent Form(s) (ICF);
4. Is scheduled for surgery that is expected to last less than 3 hours;
5. Is scheduled for any type of surgery where a single-dose perioperative cefazolin prophylaxis is appropriate.

Exclusion Criteria:

1. If female, is pregnant or lactating/breastfeeding.
2. If female that is of childbearing potential and sexually active, and is not using an effective method of birth control, e.g., oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or have a partner with a vasectomy.
3. Has a history of renal impairment -- Subject has an eGFR of <80 mL/min/1.73m2 performed at Screening as calculated by the following equation: 186 x (Creatinine/88.4)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if black) (FDA Guidance for Industry Pharmacokinetics in Patients with Impaired Renal Function)
4. Has a known allergy or hypersensitivity to β lactam/cephalosporin antibiotics, corn products, or dextrose-containing products or solutions, or any of the other ingredients of Cefazolin for Injection United States Pharmacopeia (USP) and Dextrose Injection USP in DUPLEX.
5. Has a result of any laboratory test (or repeat test, if done), obtained as standard of care, that is outside the normal limit of the site's laboratory reference range AND is considered by the investigator to be clinically significant.
6. Has had a recent (within 14 days prior to the planned surgery) administration of cefazolin.
7. Has had administration of any medication (e.g., prescription, herbal, over-the-counter medication[s] or dietary supplements) known to interact with cefazolin within 5 days prior to the study treatment administration.
8. Has a known history of human immunodeficiency virus, hepatitis B, or hepatitis C infection.
9. Has a current history of medical condition(s), which in the opinion of the investigator, would interfere with the evaluation of the study treatment.
10. Has a known history of organ transplant.
11. Has a clinically relevant disease/dysfunction of or a history of severe cardiac, pulmonary or hepatic disease.
12. Is undergoing any cardiovascular procedure including, but not limited to, major cardiac surgery, cardiac catheterizations (including electrophysiology studies), ablations, automatic implantable cardioverter-defibrillator (AICD), and pacemaker.
13. Has received any other investigational drug/device within 30 days prior to the study treatment administration.
14. Has any planned medical intervention or personal event that might interfere with ability to comply with the study requirements.
15. The subject has any condition that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the data.
16. Is unable or unwilling to adhere to the study-specified procedures and restrictions.
17. Is an employee of the Sponsor, Investigator or study-center, has direct involvement in the study or other studies under the direction of that Investigator or study-center, or is a family member of the employees or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - IACT Health - Roswell - IACT - HyperCore - PPDS, Columbus, Georgia
  - Hightower Clinical, LLC, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haessler D, Reverdy ME, Neidecker J, Brule P, Ninet J, Lehot JJ. Antibiotic prophylaxis with cefazolin and gentamicin in cardiac surgery for children less than ten kilograms. J Cardiothorac Vasc Anesth. 2003 Apr;17(2):221-5. doi: 10.1053/jcan.2003.51. PMID 12698406
- [Background] Kamath VH, Cheung JP, Mak KC, Wong YW, Cheung WY, Luk KD, Cheung KM. Antimicrobial prophylaxis to prevent surgical site infection in adolescent idiopathic scoliosis patients undergoing posterior spinal fusion: 2 doses versus antibiotics till drain removal. Eur Spine J. 2016 Oct;25(10):3242-3248. doi: 10.1007/s00586-016-4491-7. Epub 2016 Mar 12. PMID 26971263
- [Background] Khan AJ. Clinical and laboratory evaluation of cefazolin: a new cephalosporin antibiotic in pediatric patients. Curr Ther Res Clin Exp. 1973 Oct;15(10):727-33. No abstract available. PMID 4201317
- [Background] Koshida R, Nakashima E, Ichimura F, Nakano O, Watanabe R, Taniguchi N, Tsuji A. Comparative distribution kinetics of cefazolin and tobramycin in children. J Pharmacobiodyn. 1987 Sep;10(9):436-42. doi: 10.1248/bpb1978.10.436. PMID 3437384
- [Background] Lee KR, Ring JC, Leggiadro RJ. Prophylactic antibiotic use in pediatric cardiovascular surgery: a survey of current practice. Pediatr Infect Dis J. 1995 Apr;14(4):267-9. doi: 10.1097/00006454-199504000-00004. PMID 7603806
- [Background] Leggett JE, Fantin B, Ebert S, Totsuka K, Vogelman B, Calame W, Mattie H, Craig WA. Comparative antibiotic dose-effect relations at several dosing intervals in murine pneumonitis and thigh-infection models. J Infect Dis. 1989 Feb;159(2):281-92. doi: 10.1093/infdis/159.2.281. PMID 2644371
- [Background] Maher KO, VanDerElzen K, Bove EL, Mosca RS, Chenoweth CE, Kulik TJ. A retrospective review of three antibiotic prophylaxis regimens for pediatric cardiac surgical patients. Ann Thorac Surg. 2002 Oct;74(4):1195-200. doi: 10.1016/s0003-4975(02)03893-6. PMID 12400768
- [Background] Rodgers GL, Fisher MC, Lo A, Cresswell A, Long SS. Study of antibiotic prophylaxis during burn wound debridement in children. J Burn Care Rehabil. 1997 Jul-Aug;18(4):342-6. doi: 10.1097/00004630-199707000-00012. PMID 9261702
- [Background] Ross S, Rodriguez W, Khan W. The cephalosporin antibiotics in pediatric practice. South Med J. 1977 Jul;70(7):855-61. doi: 10.1097/00007611-197707000-00026. PMID 877649
- [Background] Schmitz ML, Blumer JL, Cetnarowski W, Rubino CM. Determination of appropriate weight-based cutoffs for empiric cefazolin dosing using data from a phase 1 pharmacokinetics and safety study of cefazolin administered for surgical prophylaxis in pediatric patients aged 10 to 12 years. Antimicrob Agents Chemother. 2015 Jul;59(7):4173-80. doi: 10.1128/AAC.00082-15. Epub 2015 May 4. PMID 25941220
- [Background] Schmitz ML, Rubino CM, Onufrak NJ, Martinez DV, Licursi D, Karpf A, Cetnarowski W. Pharmacokinetics and Optimal Dose Selection of Cefazolin for Surgical Prophylaxis of Pediatric Patients. J Clin Pharmacol. 2021 May;61(5):666-676. doi: 10.1002/jcph.1785. Epub 2020 Dec 9. PMID 33202066
- See also: Nahata MC, Winters CB, Powell DA. Variation in prophylactic antibiotic use in pediatric orthopedic surgery. Drug Intell Clin Pharm. 1985;19(11):834-6 — https://pubmed.ncbi.nlm.nih.gov/2998718/
- See also: Nahata MC, Durrell DE, Ginn-Pease ME, et al. Pharmacokinetics and tissue concentrations of cefazolin in pediatric patients undergoing gastrointestinal surgery. Eur J Drug Metab Pharmacokinet. 1991;16(1):49-52 — https://pubmed.ncbi.nlm.nih.gov/1936061/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no pre-assignment activities for this study.
Period: Overall Study
Arm/Group | Cefazolin 3gm Injection
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (16.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Baseline Weight [Mean (Standard Deviation); unit: kg] | 134.82 (8.133)

OUTCOME MEASURES:

1. Primary Outcome: Cefazolin Plasma Concentration Following Infusion
Description: Concentrations will be determined through analysis of 5 blood samples drawn at 0.5 (end of infusion), 1, 2, 4, and 8 hours after the start of study drug infusion.
Time Frame: 8 hours
Population: Only one (1) subject agreed to the 8-hour PK blood sample.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
ug/mL
  0.5 hours post infusion | 491 (702)
  1 hour post infusion | 117 (25.8)
  2 hours post infusion | 99.7 (21.6)
  4 hours post infusion | 57.9 (34.4)
  8 hours post infusion: number analyzed (Participants) | 1
  8 hours post infusion | 18.4 (NA) — Cannot perform STD on a single data point

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety] According to Study Protocol
Description: Safety will be assessed by monitoring adverse events (AEs), physical examination, vital signs, and clinical laboratory tests.
Time Frame: 2 days with optional visit on Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
Participants | 0

3. Secondary Outcome: Hematology: Hemoglobin (Hb)
Description: gm/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
gm/L
  Baseline | 138.5 (18.88)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 129.8 (8.93)

4. Secondary Outcome: Hematology: Hematocrit (Hct)
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
ratio
  Baseline | 0.4733 (0.08105)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 0.4066 (0.06986)

5. Secondary Outcome: Hematology: Mean Corpuscular Volume (MCV)
Description: fL
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Error); unit: fL
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
fL
  Baseline | 98.33 (10.655)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 94.98 (9.976)

6. Secondary Outcome: Hematology: Mean Corpuscular Hemoglobin (MCH)
Description: pg
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
pg
  Baseline | 28.93 (3.085)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 30.20 (0.574)

7. Secondary Outcome: Hematology: Mean Corpuscular Hemoglobin Concentration
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol/L
  Baseline | 295.1 (26.28)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 323.2 (29.99)

8. Secondary Outcome: Hematology: Platelet Count
Description: platelets / L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
10^9 platelets/L
  Baseline | 315.8 (80.08)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 236.0 (48.66)

9. Secondary Outcome: Hematology: RBC
Description: cells/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: 10^12 cells / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
10^12 cells / L
  Baseline | 4.811 (0.6083)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 4.294 (0.2875)

10. Secondary Outcome: Hematology: WBC
Description: cells/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: 10^9 cells / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
10^9 cells / L
  Baseline | 7.778 (1.6936)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 11.170 (6.4876)

11. Secondary Outcome: Clinical Chemistry: Sodium
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: mmol / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol / L
  Baseline | 140.6 (2.27)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 138.8 (1.72)

12. Secondary Outcome: Clinical Chemistry: Potassium
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 7 subjects
Measure: Mean (Standard Deviation); unit: mmol / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol / L
  Baseline | 4.32 (0.463)
  Day 2 Discharge: number analyzed (Participants) | 7
  Day 2 Discharge | 3.99 (0.776)

13. Secondary Outcome: Clinical Chemistry: Chloride
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: mmol / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol / L
  Baseline | 103.3 (3.89)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 105.5 (5.39)

14. Secondary Outcome: Clinical Chemistry: CO2 (Bicarbonate)
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: mmol / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol / L
  Baseline | 22.7 (4.10)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 22.5 (6.50)

15. Secondary Outcome: Clinical Chemistry: Glucose
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: mmol / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol / L
  Baseline | 6.36 (2.91)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 7.71 (2.24)

16. Secondary Outcome: Clinical Chemistry: ALT
Description: IU/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: IU / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
IU / L
  Baseline | 21.1 (8.35)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 28.2 (8.35)

17. Secondary Outcome: Clinical Chemistry: AST
Description: IU/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: IU / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
IU / L
  Baseline | 19.6 (5.81)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 39.0 (30.25)

18. Secondary Outcome: Clinical Chemistry: Creatine Phosphokinase (CPK)
Description: ukat / L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: ukat / L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
ukat / L
  Baseline | 2.73 (4.68)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 3.76 (3.40)

19. Secondary Outcome: Clinical Chemistry: Lactic Acid Dehydrogenase (LDH)
Description: IU/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 5 subjects
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
IU/L
  Baseline | 238.5 (68.99)
  Day 2 Discharge: number analyzed (Participants) | 5
  Day 2 Discharge | 216.8 (59.49)

20. Secondary Outcome: Clinical Chemistry: Albumin
Description: g/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
g/L
  Baseline | 39.8 (3.71)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 38.0 (4.69)

21. Secondary Outcome: Clinical Chemistry: Alkaline Phosphatase
Description: IU/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
IU/L
  Baseline | 83.08 (19.91)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 78.58 (37.15)

22. Secondary Outcome: Clinical Chemistry: Uric Acid
Description: umol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
umol/L
  Baseline | 334.7 (110.5)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 316.4 (128.8)

23. Secondary Outcome: Clinical Chemistry: Calcium
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 7 subjects
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol/L
  Baseline | 2.24 (0.106)
  Day 2 Discharge: number analyzed (Participants) | 7
  Day 2 Discharge | 2.11 (0.075)

24. Secondary Outcome: Clinical Chemistry: Phosphate
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol/L
  Baseline | 1.11 (0.29)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 1.10 (0.28)

25. Secondary Outcome: Clinical Chemistry: Total Protein
Description: g/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
g/L
  Baseline | 66.1 (3.58)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 67.2 (2.99)

26. Secondary Outcome: Clinical Chemistry: Total Bilirubin
Description: micro-mol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: micro-mol/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 9
micro-mol/L
  Baseline | 7.65 (4.17)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 7.30 (4.70)

27. Secondary Outcome: Clinical Chemistry: Blood Urea Nitrogen
Description: mmol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mmol/L
  Baseline | 6.64 (2.40)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 5.63 (1.68)

28. Secondary Outcome: Clinical Chemistry: Creatinine
Description: micro-mol/L
Time Frame: 2 days with optional visit on Day 8
Population: Medical staff only obtained clinical labs from 6 subjects
Measure: Mean (Standard Deviation); unit: Umol/L
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
Umol/L
  Baseline | 79.4 (27.5)
  Day 2 Discharge: number analyzed (Participants) | 6
  Day 2 Discharge | 68.46 (17.56)

29. Secondary Outcome: Vital Signs: Temperature
Description: Degree centigrade
Time Frame: Baseline; post-infusion at 30-minutes, 2-hours, 4-hours, and 8-hours; post-surgery
Population: Medical staff only obtained temperature from 2 subjects at the 8-hour post-infusion timepoint
Measure: Mean (Standard Deviation); unit: degrees centrigrade
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
degrees centrigrade
  Baseline | 36.5 (0.41)
  Post-Infusion, 30-min | 36.6 (0.32)
  Post-Infusion, 2-hr | 36.6 (0.31)
  Post-Infusion, 4-hr | 36.5 (0.20)
  Post-Infusion, 8-hr: number analyzed (Participants) | 2
  Post-Infusion, 8-hr | 36.8 (0.23)
  End of Surgery | 36.4 (0.28)

30. Secondary Outcome: Vital Signs: Blood Pressure (Systolic)
Description: mm Hg
Time Frame: Baseline; post-infusion at 30-minutes, 2-hours, 4-hours, and 8-hours; post-surgery
Population: Medical staff only obtained BP from 2 subjects at the 8-hour post-infusion timepoint
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mm Hg
  Baseline | 139.8 (17.8)
  Post-Infusion, 30-min | 127.9 (17.3)
  Post-Infusion, 2-hr | 128.4 (28.2)
  Post-Infusion, 4-hr | 133.9 (16.1)
  Post-Infusion, 8-hr: number analyzed (Participants) | 2
  Post-Infusion, 8-hr | 137.5 (24.8)
  End of Surgery | 139.3 (23.4)

31. Secondary Outcome: Vital Signs: Heart Rate
Description: Beats per minute
Time Frame: Baseline; post-infusion at 30-minutes, 2-hours, 4-hours, and 8-hours; post-surgery
Population: Medical staff only obtained temperature from 2 subjects at the 8-hour post-infusion timepoint
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
beats per minute
  Baseline | 79.8 (17.1)
  Post-Infusion, 30-min | 76.2 (14.2)
  Post-Infusion, 2-hr | 79.8 (15.3)
  Post-Infusion, 4-hr | 77.9 (11.6)
  Post-Infusion, 8-hr: number analyzed (Participants) | 2
  Post-Infusion, 8-hr | 80.5 (24.8)
  End of Surgery | 78.8 (12.6)

32. Secondary Outcome: Vital Signs: Respiratory Rate
Description: Breaths per minute
Time Frame: Baseline; post-infusion at 30-minutes, 2-hours, 4-hours, and 8-hours; post-surgery
Population: Medical staff only obtained temperature from 2 subjects at the 8-hour post-infusion timepoint
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
Breaths per minute
  Baseline | 17.2 (2.12)
  Post-Infusion, 30-min | 16.2 (2.69)
  Post-Infusion, 2-hr | 16.8 (4.20)
  Post-Infusion, 4-hr | 16.2 (1.47)
  Post-Infusion, 8-hr: number analyzed (Participants) | 2
  Post-Infusion, 8-hr | 17.0 (1.41)
  End of Surgery | 16.5 (4.12)

33. Secondary Outcome: Vital Signs: Weight
Description: kg
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
kg | 134.8 (8.13)

34. Secondary Outcome: Vital Signs: Height
Description: cm
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
cm | 173.4 (9.62)

35. Secondary Outcome: Vital Signs: BMI
Description: kg/cm^2
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
kg/cm^2 | 45.13 (4.84)

36. Secondary Outcome: ECG: PR Interval
Description: msec
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
msec
  Baseline | 163.8 (44.08)
  Day 2 Discharge | 154.2 (14.41)

37. Secondary Outcome: ECG: QRS Duration
Description: msec
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
msec
  Baseline | 84.0 (10.12)
  Day 2 Discharge | 90.2 (9.44)

38. Secondary Outcome: ECG: QT Interval
Description: msec
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
msec
  Baseline | 377.1 (41.19)
  Day 2 Discharge | 398.3 (35.52)

39. Secondary Outcome: Urine Pregnancy Test
Description: (If appropriate) If positive, a confirmatory serum test will be performed.
Time Frame: Baseline
Population: Pregnancy was an exclusionary criteria. All women enrolled where either post-menopausal or had a negative pregnancy test.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 7
Participants | 7

40. Secondary Outcome: Vital Signs: Blood Pressure (Diastolic)
Description: mm Hg
Time Frame: Baseline; post-infusion at 30-minutes, 2-hours, 4-hours, and 8-hours; post-surgery
Population: Medical staff only obtained BP from 2 subjects at the 8-hour post-infusion timepoint
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cefazolin 3gm Injection
Number analyzed (Participants) | 12
mm Hg
  Baseline | 80.0 (11.2)
  Post-Infusion, 30-min | 77.7 (8.49)
  Post-Infusion, 2-hr | 76.8 (17.6)
  Post-Infusion, 4-hr | 76.8 (11.5)
  Post-Infusion, 8-hr: number analyzed (Participants) | 2
  Post-Infusion, 8-hr | 77.0 (14.1)
  End of Surgery | 81.2 (12.6)

ADVERSE EVENTS:
Time Frame: Data were collected from signing of consent through the follow-up visit on End of Study (Day 8).
Arm/Group | Cefazolin 3gm Injection
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study data may be considered for reporting or publication. Sponsor will be responsible for these activities and may work with the investigators to determine how the manuscript is written, the number and order of authors, the journal, and other related issues. The sponsor has final approval authority over all such issues.

Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, which shall be in the sponsor's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05205486/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT05205486/SAP_001.pdf